CLINICAL TRIAL: NCT01147705
Title: Allopurinol as a Possible Oxygen Sparing Agent During Exercise in Peripheral Arterial Disease
Acronym: APOSA-PAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government); British Heart Foundation (Other)
Responsible Party: Principal Investigator, Alan Robertson, Clinical Research Fellow, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009CV16; 2010-020662-23 (EudraCT Number)
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral arterial disease; Allopurinol
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allopurinol (Active Comparator): Participants will be given blinded medication and asked to take one tab/day for the first six weeks (100mg strength for two weeks then 300mg strength for four weeks) followed by two tabs/day for the remaining 18 weeks.
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): Same number of tablets and appearance as active drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol — Participants will be given blinded medication and asked to take one tab/day for the first six weeks (100mg strength for two weeks then 300mg strength for four weeks) followed by two tabs/day for the remaining 18 weeks
  Arms: Allopurinol
Drug: Placebo — Same appearance/dosing as active drug.
  Arms: Placebo

SUMMARY:
Peripheral arterial disease (PAD) is a common condition that arises due to the build up of atheroma in the arteries supplying blood to the peripheral muscles and other tissues. This imbalance between oxygen supply and demand becomes particularly apparent when patients with the condition are walking. The pain and weakness they experience (mainly in the calf but less commonly in the thigh) is known as intermittent claudication and resolves upon cessation of exercise.

It is an important disease to study as it is (i) common (est. prevalence of symptomatic intermittent claudication in Scotland of 4.5%) and (ii) those with it have a 1.6 times higher relative risk of ischaemic heart disease. These patients also have a significantly higher mortality than age-matched controls at around 12% per year.

There are two main aims of therapy - (i) to reduce the risk of cardiovascular events by way of standard secondary prevention measures (smoking cessation, anti-platelet, anti-hypertensive and cholesterol-lowering therapy, diabetic control) and (ii) to treat symptoms.

Supervised exercise therapy has been shown to be beneficial in improving walking time and distance in selected patients with leg pain from intermittent claudication with an overall increase in walking distance of approximately 150 metres at three months.

There are numerous drug treatments available for consideration in PAD patients (mainly cilostazol in the UK), but many of these have either undesirable side effects or no clear evidence of benefit. The range of increase in walking distance on cilostazol was reported to be a 50-76% increase over three months compared to 20% with placebo with some significant improvements in Quality of Life (QOL) indicators, although with a significant number of adverse effects (16% vs 8% on placebo) limiting therapy. The current cost (March 2010) is £35.31/month.

Other options for therapy include angioplasty and bypass surgery. At present these are only recommended for patients who fail to respond to medical therapy and have severely disabling symptoms (in the absence of significant exercise-limiting comorbidities).

DETAILED DESCRIPTION:
The investigators will recruit 50 patients with peripheral arterial disease for a randomised, double-blind, placebo-controlled parallel group study to see if allopurinol prolongs time to leg pain and maximum walking distance as assessed by treadmill testing and the six minute walk test. Recruitment will take place in Dundee, i.e. a single-centre trial. Treatment will last for 24 weeks.

Participants will be recruited from current and past attendees at the vascular laboratory and both the intermittent claudication clinic and other outpatient clinics at Ninewells.

Participants will be allowed to continue all their usual medication throughout. After two baseline treadmill tests, they will be randomised to either allopurinol or placebo in a parallel group study and in a double blind fashion. Each participant will be on-study for 24 weeks (which is the standard time for all PAD medical intervention trials). The ultimate dose of allopurinol will be 300 mg BD, which is the dose known to work in angina. However, for safety purposes, the initial dose will be 100 mg/day for two weeks, rising to 300 mg/day for four weeks, followed by 600 mg/day for the next 18 weeks. Participants and their bloods (UE, LFT, FBC) will be monitored at weeks 0, 6, 18 and 24 weeks and medication stopped or reduced in dose if concerns arise. If study drug dose is reduced, they will stay in study. If study drug needs to be stopped, they will stay in study in order to do an "intention to treat" analysis.

Double blind medication (allopurinol or placebo) will be prepared and packaged by Tayside Pharmaceuticals. The medication will come labelled as "Participant 1", "Participant 2", etc. and will be distributed to the participant by the research fellow according to their sequence number. The blinded treatment code will be kept by the Clinical Trials Pharmacy Department, Ninewells, who operate a 24 hour emergency unblinding facility (as necessary) and in a sealed envelope in a locked fireproof cabinet accessible by a responsible member of University of Dundee staff not directly involved in the study.

The following is the programme of visits involved in this study (list taken from the participant information sheet) -

* Visit 1 (week 0) - screening visit 1

  * Consent - answer any outstanding questions you may have and complete the consent form.
  * Measurement of blood pressure in arms and legs
  * Treadmill test
  * Blood samples
* Visit 2 (week 0) - screening visit 2

  * Treadmill test - if this is stable and similar to the previous test then you are able to continue in the study
  * Six minute walk test
  * Measurement of blood vessel 'stiffness'
  * Supply of initial study medication along with instructions.
  * Two questionnaires - Walking Impairment and Quality of Life
* Visit 3 (week 6) - progress visit

  * Check how you are doing on the medications
  * Blood samples
  * Supply of study medication for the remainder of the study
* Visit 4 (week 12) - progress visit

  * Treadmill test
  * Six minute walk test
  * Check how you are doing on the medications
  * Two questionnaires - Walking Impairment and Quality of Life
* Visit 5 (week 18) - progress visit

  * Measurement of blood vessel 'stiffness'
  * Check how you are doing on the medications
  * Blood samples
* Visit 6 (week 24) - final visit

  * Measurement of blood vessel 'stiffness'
  * Treadmill test
  * Six minute walk test
  * Measurement of blood pressure in arms and legs
  * Check how you are doing on the medications
  * Blood samples
  * Two questionnaires - Walking Impairment and Quality of Life

ELIGIBILITY:
Inclusion Criteria:

- stable peripheral arterial disease (demonstrated by having a reproducible pain free walking distance on 2 consecutive treadmill tests, i.e. less than 25% variance with the reason for termination of the treadmill test must be claudication pain only)

Exclusion Criteria:

* rest pain
* childbearing potential
* heart failure
* any other exercise limiting cardiac disease
* BP > 180/100 mHg
* eGFR < 60 ml/min
* liver disease
* malignancy
* already on allopurinol or had an adverse reaction to it
* recent marked change in symptoms or recent (in the last six months) intervention for PAD
* receiving treatment with either 6-mercaptopurine, azathioprine, warfarin, or theophylline

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Onset of claudication pain | 24 weeks
  Our primary endpoint will be the distance to onset of claudication pain at 24 weeks but we will also measure total exercise distance.

SECONDARY OUTCOMES:
Quality of life | 24 weeks
  To see if allopurinol improves quality of life in patients with PAD.
Anti-oxidant effects | 24 weeks
  To investigate the anti-oxidant effects of allopurinol of patients with PAD.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Struthers, MD FRCP, Study Director — University of Dundee; Alan J Robertson, MBChB MRCP, Principal Investigator — University of Dundee
Locations (1):
- Ninewells Hospital, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robertson AJ, Struthers AD. A Randomized Controlled Trial of Allopurinol in Patients With Peripheral Arterial Disease. Can J Cardiol. 2016 Feb;32(2):190-6. doi: 10.1016/j.cjca.2015.05.010. Epub 2015 May 19. PMID 26277090